CLINICAL TRIAL: NCT00752999
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Dose Study of R935788 in Systemic Lupus Erythematosus Patients With Active Disease
Brief Title: Efficacy and Safety Study of R935788 Tablets to Treat Systemic Lupus Erythematosus
Acronym: SOLEIL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn for business reasons before study start.
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-015; 2008-004472-50 (EudraCT Number)
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 150 mg tablet, oral, twice-a-day
  Interventions: Drug: Fostamatinib Disodium (R935788)
- B (Placebo Comparator): Placebo tablet, oral, twice-a-day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib Disodium (R935788) — 150 mg tablet, oral, twice-a-day
  Other Names: R788
  Arms: A
Drug: Placebo — Placebo tablet, oral, twice-a-day
  Arms: B

SUMMARY:
Approximately 225 patients meeting study entry requirements will be enrolled and randomized (2:1, active versus placebo superimposed on background treatment) to R788 or placebo. Patients will be followed for efficacy and safety parameters for 6 months. The investigator should taper corticosteroids if clinically warranted.

DETAILED DESCRIPTION:
This study is a multi-center, multinational, randomized, double-blind, placebo-controlled Phase II clinical trial. Study enrollment will comprise approximately 225 patients meeting study inclusion requirements. The study will be conducted at up to 80 multinational investigational sites. Eligible patients will be randomized (2:1) into one of two 6 month treatment groups. One group (approximately 150 patients) will receive R788 150 mg PO bid; the other treatment group (approximately 75 patients) will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent to participate in this study by signing an IRB/EC-approved Informed Consent Form (ICF) prior to admission to this study.
* Males and females, 18 years of age or older, with active SLE diagnosed at least 6 months prior to Day 1 dosing. Active SLE is defined as having fulfilled the ACR criteria for SLE.
* Patients of childbearing potential must be fully informed of the potential for R788 to adversely affect the fetus and, if sexually active, must agree to use an effective method of birth control during the study (oral contraceptive, mechanical barrier, long acting hormonal agent).
* The patient must otherwise be in good health as determined by the investigator on the basis of medical history, physical examination, and laboratory screening tests during the screening period.
* In the investigator's opinion, the patient has the ability to understand the nature of the study and any anticipated risks of participation, communicate satisfactorily with the investigator, and participate in and comply with the requirements of the entire protocol.

Exclusion Criteria:

* The patient has a history of, or a concurrent, clinically significant illness, medical condition or laboratory abnormality that, in the investigator's opinion, could affect the conduct of the study.
* Clinically significant or uncontrolled medical disease in any organ system, other than due to SLE.
* Background immunosuppressive therapy that has not remained stable ≤ 4 weeks prior to baseline.
* Severe active or unstable renal disease.
* Active severe neuropsychiatric SLE.
* Female patients must not be breastfeeding and must have a negative urine pregnancy test per the Schedule of Study Activities.
* The patient has a history of substance abuse, drug addiction, or alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is defined as the decrease from baseline in the SELENA-SLEDAI score at 6 months. | 6 months

SECONDARY OUTCOMES:
Composite Responder analysis defined as ≥4 points improvement in SELENA-SLEDAI and no 'Severe SLE flare' after Week 6. No worsening (≤10 mm on VAS) of Physician Global Assessment, or, no worsening of SF 36 PCS (not >-0.8) or PFI (not >2.5) | 3 and 6 months
Attainment of daily prednisone dose decrease in those patients on daily corticosteroids by 50% or to ≤ 7.5 mg prednisone (or equivalent for other corticosteroids) at 3 and 6 months. | 3 and 6 months
Decrease from baseline in SELENA-SLEDAI score at each post baseline visit. | At each post baseline visit
Attainment of improvement in SELENA-SLEDAI by ≥ 2 points at Weeks 2 and 4. | Weeks 2 and 4
Attainment of improvement in SELENA-SLEDAI by ≥ 4 points at each post baseline visit. | At each post baseline visit
Change from baseline of Physician Global Assessment by VAS over 6 months. | 6 months
Time to rescue medication. | At each post baseline visit
Time to severe SLE flare by SELENA Flare Index. | At each post baseline visit
Change from baseline in the component scores of the SF 36 at Month 3 and Month 6. | Month 3 and 6
Effects on liver function tests, clinically significant reductions in peripheral neutrophil counts, G-I adverse effects, new onset or aggravated hypertension, and other adverse effects as they may appear. | At each post baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B. Magilavy, MD, Study Director — Rigel Pharmaceuticals,Inc.